CLINICAL TRIAL: NCT05016011
Title: Phase IIb Study Assessing the Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cells for Knee Cartilage Injury
Brief Title: Efficacy of Allogeneic UCMSCs for Treating Large Defects Knee Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytopeutics Sdn. Bhd. (Industry)
Collaborators: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POD0032/CP/R
Record Dates: First submitted 2020-11-15; First posted 2021-08-23 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) (Experimental): Patients will receive 25 x 10^6 of human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) with standard treatment.
  Interventions: Biological: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs)
- Marrow cellution (standard treatment) (Active Comparator): Patients will undergo marrow cellution surgical procedure.
  Interventions: Procedure: Marrow cellution

INTERVENTIONS:
Biological: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) — Human umbilical cord-derived mesenchymal stem cells
  Other Names: Chondrocell-EX
  Arms: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs)
Procedure: Marrow cellution — Patients will undergo marrow cellution surgical procedure.
  Arms: Marrow cellution (standard treatment)

SUMMARY:
In terms of the surgical treatment of the cartilage injury, various techniques and ways are created to repair or regenerate articular surface of synovial joint following traumatic damage or degeneration of the cartilage. The option for surgical treatments based on the size and depth of the cartilage knee injury may include knee debridement, radiofrequency, drilling, microfracture, mosaicplasty, allogenic osteochondral transplantation and autologous chondrocyte transplantation. The first two techniques mentioned have been used in treating the cartilage knee injury involving the partial defects meanwhile the latter techniques have been used for Grade III and IV cartilage defects based on ICRS. However, most of the surgical options up only provide more of Type I collagen rather than Type II collagen. The available treatments are more symptomatic rather than preventive or regenerative. Stem cell has big potential in this area where it has ability to differentiate to cartilage. As allogeneic umbilical cord blood MSCs are readily available and can be administered immediately, this study therefore aims to prove the efficacy of allogeneic umbilical cord-derived mesenchymal stem cells (UC-MSCs) for treating large defects knee injury.

The study is a prospective, randomized controlled, open label, phase IIb clinical trial, involving 50 patients with large defects of cartilage injury for follow-up duration of 24 months. Patients will be assigned into 2 arms; Arm A - 25 subjects will receive Chondrocell-EX (UC-MSCs) and Arm B - 25 subject will receive marrow cellution. All patients will undergo debridement prior to receiving their assigned treatment. The patients will be assessed on KOOS, IKDC, VAS and MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 65 years.
2. Patients diagnosed to have ICRS Grade 3 or 4 cartilage lesions based on the MRI scans of the affected knee.
3. Presence of knee swelling, pain, stiffness, or knee mechanical symptoms resulting from cartilage lesions.
4. All subjects must also satisfy at least 1 of the following inclusion criteria.

   * Isolated knee articular cartilage lesion (single lesion) estimated to be ≥1.0 cm2 as demonstrated on MRI scanning.
   * Multiple knee articular cartilage lesions (multiple lesions) with at least 1 lesion estimated to be ≥1.0 cm2 as demonstrated on MRI scanning.
   * Bipolar cartilage defects demonstrated on MRI scanning with at least 1 articular surface lesion to be ≥1.0 cm2.
   * One or more cartilage defects involving the patella-femoral joint as demonstrated on MRI scanning with at least 1 lesion ≥1.0 cm2.
   * One or more cartilage defects involving the tibio-femoral joint as demonstrated on MRI scanning with at least 1 lesion ≥1.0 cm2.
   * Previously failed cartilage repair procedures (i.e., microfracture, osteochondral autograft transplantation surgery (OATS), ACI) within 6 months.

Exclusion Criteria:

1. Preoperative flexion deformity greater than 10 degrees.
2. Significant cognitive impairment, non-ambulatory status or lower extremities amputation other than toes, serious illness or medication affecting operative risk or wound healing (e.g., steroid intake, anticoagulation).
3. Patient with high co-morbidity
4. Higher risk for postsurgical (e.g., bleeding disorder or taking anticoagulants except low-dose aspirin) or postsurgical infection (e.g., taking immune-suppressants, have a severe infection or a history of serious infection).
5. Significant peripheral vascular disease of the lower limbs as indicated by absent or substantially reduced dorsalis pedis or posterior tibial pulses.
6. Contraindications to sub-chondral drilling surgery.
7. Women who are pregnant or who are not able to use contraceptives
8. Known hypersensitivity (allergy) to hyaluronate or antibodies used for postsurgical prophylaxis.
9. Infections or skin disease affecting the area of the injection site or joint.
10. Intra-articular injections of hyaluronic acid in the target knee within the past 6 months before screening.
11. Intra-articular injections of corticosteroids in the target knee within the past 3 months before screening.
12. In the opinion of the investigators, the subjects have difficulty understanding or complying with the protocol procedures or requirements including follow up.
13. In the opinion of the investigators, the subject has any medical, psychiatric, or other condition for which the study would pose particular safety risks and/or unfavorably affect the risk-benefit balance of participation.
14. Presence of metallic implants, clips, or devices in the brain, eye, or spinal canal or implanted devices that are magnetically programmed that may affect the ability to perform MRI MOCART scoring.
15. Significant knee malalignment, varus or valgus deformity with more than 10 degrees, or instability associated with ligamentous knee injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Recording of Adverse Events and Serious Adverse Events | 24 months
International Knee Documentation Committee (IKDC) score | 24 months
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 24 months
Visual Analog Score (VAS) | 24 months
Immunohistochemistry (IHC) | 12 months
  IHC staining for generated cartilage

CONTACTS AND LOCATIONS:
Overall Officials: Badrul Akmal Hisham Md Yusoff, Principal Investigator — Hospital Canselor Tuanku Muhriz Universiti Kebangsaan Malaysia (HCTM-UKM)
Locations (1):
- Hospital Canselor Tuanku Muhriz Universiti Kebangsaan Malaysia (HCTM-UKM), Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No